CLINICAL TRIAL: NCT03930862
Title: Comparison of Muscle Activity and Patients Satisfaction on Implants Supported Overdenture Using Ball and Socket Versus Locator Attachment
Brief Title: Ball and Socket Versus Locator Attachment Retained Implant Overdentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lamees Hosam Ramadan (Other)
Responsible Party: Sponsor-Investigator, Lamees Hosam Ramadan, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Muscle activity
Record Dates: First submitted 2019-04-05; First posted 2019-04-29 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Complete Edentulism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ball and socket (Active Comparator): It is an attachment retaining implant overdentures to increase retention and stability of the denture
  Interventions: Device: Locator Attachment (positioner)
- Locator attachment (Experimental): attachment retaining implant overdentures
  Interventions: Device: Locator Attachment (positioner)

INTERVENTIONS:
Device: Locator Attachment (positioner) — intra oral attachment

SUMMARY:
Will the use of locator attachment influence the muscle efficacy when compared to ball and socket attachment in mandibular implant overdenture? '

DETAILED DESCRIPTION:
In this study we will use a two different types of attachments in implants overdenture in mandibular completely edentulous patients to increase the retention and stability of the denture and this can be recognized by record the masticatory function of the muscles of the mandibular jaw.

ELIGIBILITY:
Inclusion Criteria:

- Upper and lower completely edentulous patients. Acceptance of the existing denture if it is good, or constructing a new one if it is defected.

Patients with adequate bone quality and quantity. Tooth extracted not less than 6 month.

Exclusion Criteria:

1. Young patients.
2. Diseases affecting neuromuscular coordination.
3. TMJ diseases.
4. Soft tissue abnormalities.
5. Bony exostosis.
6. Parathyroid dysfunction
7. uncontrolled Diabetes
8. Radiotherapy to the neck or head
9. Pregnancy.
10. Drug and alcohol dependency.
11. Smokers.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Activity | 6 month
  Digital Electromyogram

SECONDARY OUTCOMES:
Patient Satisfaction: questionnaire | 6 month
  questionnaire from zero to 10 where zero is completely unsatisfied and 10 is highly satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Nada Sherine, PhD, Study Director — Lecturer of Prosthdontics

IPD SHARING:
Plan to Share IPD: No